CLINICAL TRIAL: NCT01268384
Title: Phase II Study of Fixed Dose Rate Gemcitabine Plus Capecitabine in Locally Advanced Pancreatic Cancer
Brief Title: Neoadjuvant FDR GX in Locally Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, JLee, Associate professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APBCC_01
Record Dates: First submitted 2010-12-29; First posted 2010-12-30 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; neoadjuvant chemotherapy; gemcitabine; capecitabine
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Capecitabine; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FDR_GX (Experimental): Fixed dose rate gemcitabine plus capecitabine every 3 weeks for 3-9 cycles
  Interventions: Drug: Gemcitabine plus Capecitabine

INTERVENTIONS:
Drug: Gemcitabine plus Capecitabine — Gemcitabine 1,250 mg/m2 mixed with 0.9% saline 500 ml i.v. for 10 mg/m2/min on D1 and D8 Capecitabine 950 mg/m2 b.i.d. po from D1 to D14 every 21 days
  Other Names: Neoadjuvant chemotherapy; GemCap

SUMMARY:
The rationale for phase II trial of neoadjuvant fixed dose rate gemcitabine plus capecitabine for patients with LAPC includes the following: First, obtaining a sufficient tumor down-staging to procure R0/R1 resection, reported to be one of the most significant prognostic factors for survival; second, providing an observation period to exclude from surgery those patients with rapidly progressive disease there by to help select patients for surgery who have the greatest likelihood of a favorable postoperative outcome; third, eliminating micrometastatic disease, that is likely present in most patients, earlier than adjuvant setting and preventing post-surgical growth spurts; fourth, adjuvant therapy given in the neoadjuvant setting is better tolerated, as the patient has not recently undergone a major operation; and the last, the lack of widely accepted optimal preoperative or palliative approach in patients with LAPC, the majority of whom may not be operated on.

The primary goal is to determine the R0 resection rate of the neoadjuvant fixed dose rate (FDR) gemcitabine-capecitabine combination chemotherapy in patients with borderline resectable or unresectable locally advanced pancreatic adenocarcinoma.

The secondary goals are to assess progression-free survival (PFS) and OS (overall survival) in these patients and to assess adverse events of these neoadjuvant treatments.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented pancreatic adenocarcinoma
* Clinical T3 or T4 tumor according to AJCC staging system
* Tumors considered as borderline resectable or unresectable disease assessed by multidisciplinary team including pancreatic surgeon, gastroenterologist specializing in pancreas, medical oncologist, and radiation oncologist
* Age 18 years or older
* ECOG performance status 2 or less
* Adequate organ function

  * Adequate bone marrow function (WBCs> 3,500/µL, absolute neutrophil count [ANC]> 1,500/µL, hemoglobin > 9.0 g/dL, and platelets > 100,000/µL)
  * Adequate kidney function (creatinine < 1.5 mg/dL)
  * Adequate liver function (bilirubin < 1.5 mg/dL [<2.5 mg/dL for patients with obstructive jaundice due to pancreatic cancer with adequate decompression], transaminases levels < 3 times the upper normal limit)
* Patients must not have psychological, familial, sociological or geographical conditions which do not permit medical follow-up and compliance with this study
* Women of childbearing potential must have a negative pregnancy test on admission. Post-menopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential. Men and women of reproductive potential must have agreed to use an effective method of contraception while on treatment and for 6 months after study treatment
* The patient must be able to understand the study and has given written informed consent to participate in the study

Exclusion Criteria:

* Other tumor type than adenocarcinoma
* Evidence of gastrointestinal bleeding or obstruction
* Presence of the clinically relevant ascites or distant metastases
* Past or concurrent history of malignant neoplasm, except for curatively treated non-melanoma skin cancer or in situ carcinoma of the cervix uteri
* Pregnant or lactating women, women of childbearing potential not employing adequate contraception
* Hypersensitivity to any of the study drugs or ingredients
* Other serious illness or medical conditions

  * Unstable cardiac disease despite treatment, myocardial infarction within 6 months prior to study entry
  * History of significant neurologic or psychiatric disorders including dementia or seizures
  * Active uncontrolled infection
  * Pre-existing clinically significant diarrhea
  * Active peptic ulcer
  * Severe hypercalcemia of 12 mg/dL uncontrolled with bisphosphonates
  * Active disseminated intravascular coagulation
  * Other serious underlying medical conditions which could impair the ability of the patient to participate in the study
* Concomitant or administration of any other experimental drug under investigation within 3 weeks before the study
* Concomitant chemotherapy, hormonal therapy, or immunotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2006-04; Primary Completion 2010-07 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
R0 resection rate | 6 months
  Microscopic complete resection rate after neoadjuvant chemotherapy

SECONDARY OUTCOMES:
Adverse events associated with neoadjuvant chemotherapy | 6 months
  NCI CTCAE v.3.0 based AEs
Overall survival | 2 years
  Overall survival after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Lyun Lee, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea